CLINICAL TRIAL: NCT02387229
Title: Blinded Randomized Trial of Anticoagulation to Prevent Ischemic Stroke and Neurocognitive Impairment in AF (BRAIN-AF)
Brief Title: Blinded Randomized Trial of Anticoagulation to Prevent Ischemic Stroke and Neurocognitive Impairment in AF
Acronym: BRAIN-AF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Consensus BRAIN-AF Executive Steering Committee to terminate.
Sponsor: Montreal Heart Institute (Other)
Collaborators: Canadian Stroke Prevention Intervention Network (Other); The Montreal Health Innovations Coordinating Center (MHICC) (Other); Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry); Montreal Heart Institute Foundation (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Hewitt Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BRAIN-001
Record Dates: First submitted 2015-02-26; First posted 2015-03-12 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: ATRIAL FIBRILLATION
Keywords: Atrial Fibrillation; Stroke; Neurocognitive decline; Rivaroxaban; Acetylsalicylic acid; Anticoagulation; Montreal Cognitive Assesssment (MoCA); Mini-Mental State Examination (MMSE)
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Active Comparator): Rivaroxaban 15 mg, orally, once daily, preferably at the same time of the day throughout the study.
  Interventions: Drug: Rivaroxaban
- standard of care (Active Comparator): standard of care
  Interventions: Other: standard of care

INTERVENTIONS:
Drug: Rivaroxaban — 15 mg
  Other Names: Xarelto
  Arms: Rivaroxaban
Other: standard of care
  Arms: standard of care

SUMMARY:
This is a prospective, multicenter, randomized, double-blinded clinical trial exploring the efficacy and safety of rivaroxaban as compared to standard of care in reducing stroke, transient ischemic attack (TIA) and neurocognitive decline, in subjects with non-valvular AF and with low risk of stroke.

DETAILED DESCRIPTION:
Subjects who qualify will be approached and those consenting will be enrolled to undergo a baseline evaluation. Subjects without a clinical diagnosis of dementia and with a Mini Mental State Examination score (MMSE) score ≥ 25 will undergo neurocognitive assessment (MoCA), psychosocial and QoL assessment before randomization.

Subjects will undergo regular visits (in-clinic, and/or by phone, or video conferencing) every 6 months during the treatment period. Subjects will take either rivaroxaban 15 mg or standard of care.

An independent clinical event committee will classify all endpoint events. An independent Data Safety Monitoring Committee (DSMC) was established to monitor the progress of the study and assure the safety of subjects enrolled in the trial.

ELIGIBILITY:
For entry into the study, the following criteria must be met:

Inclusion Criteria:

* Age at consent ≥30 to ≤62 years;
* Non-valvular atrial fibrillation (paroxysmal, persistent or permanent) documented by any electrical tracing or any device (i.e. routine 12-lead electrocardiogram, Holter monitor [continuous ECG recording] rhythm strip, intracardiac electrogram, or pacemaker or implantable cardiac defibrillator interrogation of at least 30 s, transcutaneous monitoring or other) in the last 2 years;
* Low risk of stroke as defined by the absence of all of the following:

  i. Prior stroke or Transient Ischemic Attack, ii. Hypertension, iii. Diabetes mellitus, iv. Congestive heart failure (New York Heart Association class II or higher at the time of enrolment or a known left ventricular ejection fraction <35%);
* Signed informed consent

For entry into the study, none of the following criteria MUST be met

Exclusion Criteria:

* Known diagnosis of dementia;
* MMSE score <25;
* Valvular AF [mechanical heart valve, moderate to severe mitral stenosis (rheumatic or non rheumatic), or hypertrophic cardiomyopathy];
* Other indication for antiplatelet therapy or anticoagulation;
* History of GI bleeding;
* Conditions associated with an increased risk of bleeding described as follows:

  1. Major surgery within the previous month;
  2. Planned surgery or intervention within the next 3 months;
  3. History of intracranial, intraocular, spinal, retroperitoneal or a traumatic intra-articular bleeding;
  4. Symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30 days;
  5. Haemorrhagic disorder or bleeding diathesis;
  6. Fibrinolytic agents within 48 hours of study entry;
  7. Recent malignancy or radiation therapy (within 6 months from the time of enrolment) and not expected to survive 3 years;
* Reversible cause of AF (e.g. cardiac surgery, pulmonary embolism, untreated hyperthyroidism);
* Absence of recurrence of AF 3 months after AF ablation;
* Severe renal impairment (creatinine clearance 30 mL/min or less);
* Active infective endocarditis;
* Active liver disease (e.g. acute clinical hepatitis, chronic active hepatitis, cirrhosis), or Alanine Transaminase (ALT) >3 times the upper limit of normal;
* Women who are pregnant or of childbearing potential not using a medically acceptable form of contraception throughout the study;
* Women who are breastfeeding;
* Anemia or thrombocytopenia (according to the normal range values of the local laboratory);
* Participation in another study involving an investigational drug (under development) at the same time or within 30 days of randomization;
* Subjects considered unreliable, or having a life expectancy of less than 3 years or having any condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g. drug addiction, alcohol abuse);
* History of allergic reaction to rivaroxaban.
* History of allergic reaction, in the absence of desensitization to acetylsalicylic acid in patients with vascular disease.

Ages: 30 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1238 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of stroke, TIA and neurocognitive decline. Neurocognitive decline is defined by a decrease in the MoCA score greater than or equal to 2 at any follow-up visit from baseline. | estimated up to 84 months
  From date of randomization until the date of first documented occurrence of any component of the composite, assessed up to the end of the study

SECONDARY OUTCOMES:
Death (total and cardiovascular) | estimated up to 84 months
  From date of randomization until the date of first documented death (total and cardiovascular), assessed up to the end of the study
Composite including stroke/transient ischemic attack (TIA) and systemic embolic events | estimated up to 84 months
  From date of randomization until the date of first documented composite including stroke/transient ischemic attack (TIA) and systemic embolic events, assessed up to the end of the study
Neurocognitive decline | estimated up to 84 months
  From date of randomization until the date of first documented neurocognitive decline, assessed up to the end of the study. First occurrence of decrease in MoCA score ≥2 at any follow up visit from baseline.
Hospitalization for cardiovascular (myocardial infarction, heart failure, AF, stroke or unstable angina or other cardiovascular events) or bleeding event | estimated up to 84 months
  From date of randomization until the date of first documented hospitalization for cardiovascular (myocardial infarction, heart failure, AF, stroke, other cardiovascular events or bleeding event, assessed up to the end of the study. Hospitalization is defined as an admission to an inpatient unit or a visit to an emergency department that results in at least a 24 hour stay

OTHER OUTCOMES:
Major clinical bleeding event | estimated up to 84 months
  From date of randomization until the date of first documented major clinical bleeding event, assessed up to the end of the study. First occurrence of bleeding events consider as major or requiring hospitalization. Bleeding will be defined in accordance with the International Society on Thrombosis and Haemostasis (ISTH).

CONTACTS AND LOCATIONS:
Overall Officials: Lena Rivard, MD, Principal Investigator — Montreal Heart Institute; Sophie Tanguay, M.Sc., Study Director — Montreal health Innovations Coordinating Centre
Locations (40):
- Canada (40):
  - CardiAi Inc., Calgary, Alberta
  - Libin Cardiovascular Institute of Alberta, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Office of Dr. TunZan Maung, MD, Abbotsford, British Columbia
  - North Shore Heart Center, North Vancouver, British Columbia
  - Vancouver General Hospital/UBC, Vancouver, British Columbia
  - Cardio 1, Winnipeg, Manitoba
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Dr. Georges-L - Dumont University Hospital Center, Moncton, New Brunswick
  - QEll Health Sciences Center-Halifax Infirmary, Halifax, Nova Scotia
  - Western University - London Health Sciences Centre, London, Onatrio
  - PACE (Partners in Advanced Cardiac Evaluation), Newmarket, Onatrio
  - Oakville Cardiovascular Research LP, Oakville, Onatrio
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - Vizel Cardiac Research, Cambridge, Ontario
  - Hamilton Health Sciences - General Site, Hamilton, Ontario
  - McMaster University, Hamilton, Ontario
  - Cardiology Clinic, Kitchener, Ontario
  - St. Mary's general Hospital, Kitchener, Ontario
  - One Heart Care, Mississauga, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Viacar Recherche Clinique Inc., Brossard, Quebec
  - CIUSSS du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - CIUSSS de l'Estrie-CHUS-Centre Haute-Yamaska (Hopital de Granby), Granby, Quebec
  - CISSSMC-Hopital Charles-Lemoyne, Greenfield Park, Quebec
  - Viacar Recherche Clinique Inc., Greenfield Park, Quebec
  - Hopital de la Cite-de-la-Sante, Laval, Quebec
  - Clinique Cardiologie de Levis, Lévis, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM, Montreal, Quebec
  - Hopital du Sacre Coeur de Montreal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - CISSS BSL-Hopital de Rimouski, Rimouski, Quebec
  - CISSS des Laurentides-Unite de recherche clinique, Saint-Jérôme, Quebec
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec
  - CISSS de Lanaudiere-Hopital Pierre-Le Gardeur, Terrebonne, Quebec
  - CIUSSS MCQ CHAUR- Centre Hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec
  - CHU de Quebec-Universite Laval/Hotel Dieu de Quebec, Québec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec

REFERENCES:
- [Derived] Rivard L, Khairy P, Talajic M, Tardif JC, Healey JS, Black SE, Andrade JG, Field TS, Nault I, Bherer L, Massoud F, Nattel S, Lanthier S, Racine N, Roux JF, Greiss I, Macle L, Guerra PG, Tadros R, Mayrand H, Gosselin G, Conen D, Bocti C, Chayer C, Deschaintre Y, Sandhu RK, Manlucu J, Khaykin Y, Verma A, Mondesert B, Dyrda K, Cadrin-Tourigny J, Thibault B, Raymond-Paquin A, Aguilar M, Brouillette J, Roussin A, Robillard A, Tremblay-Gravel M, David LP, Cossette M, Parkash R, Guertin MC, Roy D; BRAIN-AF investigators. Anticoagulation to prevent ischemic stroke and neurocognitive impairment in atrial fibrillation: the BRAIN-AF randomized clinical trial. Nat Med. 2026 Jan;32(1):297-305. doi: 10.1038/s41591-025-04101-y. Epub 2026 Jan 7. PMID 41501492
- [Derived] Rivard L, Khairy P, Talajic M, Tardif JC, Nattel S, Bherer L, Black S, Healey J, Lanthier S, Andrade J, Massoud F, Nault I, Guertin MC, Dorian P, Kouz S, Essebag V, Ellenbogen KA, Wyse G, Racine N, Macle L, Mondesert B, Dyrda K, Tadros R, Guerra P, Thibault B, Cadrin-Tourigny J, Dubuc M, Roux JF, Mayrand H, Greiss I, Roy D. Blinded Randomized Trial of Anticoagulation to Prevent Ischemic Stroke and Neurocognitive Impairment in Atrial Fibrillation (BRAIN-AF): Methods and Design. Can J Cardiol. 2019 Aug;35(8):1069-1077. doi: 10.1016/j.cjca.2019.04.022. Epub 2019 May 7. PMID 31376908